CLINICAL TRIAL: NCT03299777
Title: Correlation Between Changes in Liver Stiffness and Preeclampsia as Shown by Fibroscan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0036-17-NHR
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: A control group will consist 100 normotensive women with normal pregnancy outcomes who were admitted to our fetal-maternal unit during the same period
- Preeclampsia group: All patients diagnosed with preeclampsia will undergo the fibroscan test.

SUMMARY:
Compare the Fibroscan results of preeclamptic women to normal controls and to find out if the changes are reversible after labor.

Materials and Methods

DETAILED DESCRIPTION:
The purpose of the study is to compare the Fibroscan results of preeclamptic women to normal controls and to find out if the changes are reversible after labor.

Materials and Methods This prospective observational case-control study will include 50 women admitted to the fetal-maternal Unit at 24 - 41 weeks gestation and diagnosed with mild/severe preeclampsia. Preeclampsia is diagnosed as a new onset of hypertension over 140/90, at least two measurements at least four hours apart, and proteinuria (≥+1 in dipstick or >300 mg/24 hr) after 20 weeks of gestation in a previously normotensive woman.

A control group will consist 100 normotensive women with normal pregnancy outcomes who were admitted to our fetal-maternal unit during the same period. Demographic, clinical, laboratory and sonographic data for the women participating will be collected from their chart. All patients diagnosed with preeclampsia will undergo the following workup: sign and symptoms evaluation, blood pressure follow up, 24-hour protein excretion in grams per day, complete blood count, hepatic function test: AST, ALT and coagulation study, HBA1C, coagulation function test and fibrotest. The Fibroscan test will be performed by a trained hepatologist, who was blind to the women diagnosis. The fibroscan test will be done during the admission after the diagnosis of preeclampsia, after delivery and 6 weeks post-partum.

Commonly used cutoffs are >7 kPa for significant fibrosis. Statistical analysis will be performed with SPSS using Mann Whitney test. Continuous variables will be analyzed using the student's T test and categorical variables were analyzed using 2. Statistical significance was set at a P value of < 0.05. The local institutional review board approved this study.

ELIGIBILITY:
Inclusion Criteria:

- Fetal-maternal Unit at 24 - 41 weeks gestation and diagnosed with mild/severe preeclampsia

Exclusion Criteria:

* Age less then 18
* Fetal-maternal less then 24 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Materials and Methods This prospective observational case-control study will include 50 women admitted to the fetal-maternal Unit at 24 - 41 weeks gestation and diagnosed with mild/severe preeclampsia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Comparing the Fibroscan results of preeclamptic women to normal controls and to find out if the changes are reversible after labor. Fibrotic tissue differs from healthy tissue in the way it responds to excitation | 2 years
  Transient elastography is performed using transducer-induced vibrations at low frequency (50 Hz) and amplitudes. The transmitted shear waves propagate through the liver parenchyma. Pulse-echo ultrasound acquisition is used to follow the propagation of the shear wave and to measure its average speed. Results are expressed in kPa and can range from 2.5 to 75 kPa. Commonly used cutoffs in clinical settings are >7 kPa for significant fibrosis and >11 to 14 kPa for cirrhosis and CAP>270 db/m2 for significant steatosis.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Wolf, MD, Principal Investigator — Western Galilee Medical Center
Locations (1):
- Galil Medical Center, Nahariya, Israel

REFERENCES:
- [Derived] Carmiel Haggai M, Sgayer I, Bornstein J, Odeh M, Lowenstein L, Frank Wolf M. Liver stiffness and steatosis in preeclampsia as shown by transient elastography-a prospective cohort study. Am J Obstet Gynecol. 2022 Sep;227(3):515.e1-515.e9. doi: 10.1016/j.ajog.2022.04.048. Epub 2022 Apr 29. PMID 35500613